CLINICAL TRIAL: NCT03942731
Title: Resensitization Rate After Drug Provocation Test and Challenge in Eighty-three Adult Outpatients With a Distant Penicillin Allergy.
Brief Title: Penicillin Allergy Testing and Resensitization Rate
Acronym: Penicillin
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-03Obs-CHRMT
Record Dates: First submitted 2019-03-29; First posted 2019-05-08 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-03

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: 83 adult outpatients at CHR Metz-Thionville with penicillin allergy label
  Interventions: Other: Behavioral allergy testing protocol

INTERVENTIONS:
Other: Behavioral allergy testing protocol — skin tests followed by drug provocation test and skin retesting between 6 weeks and 6 months

SUMMARY:
Penicillin is one of the earliest discovered antibiotics and a drug of choice for several infections. Up to 10 to 20% of all patients in clinical trial are labeled as penicillin allergic. Most of these patients do not have a true allergy but few have had it verified. Approximately 80% of patients with IgE-mediated penicillin allergy lose their sensitivity after 10 years. Several studies have been conducted denying the risk of sensitization following negative testing of penicillin allergy. Investigators have not had the same experience and have therefore decided to conduct a retrospective study review of 83 adult outpatients with a distant penicillin allergy label and evaluate outcomes of skin retesting six weeks following Drug Provocation Test and challenge.

ELIGIBILITY:
Inclusion Criteria:

- 18 years old

Exclusion Criteria:

* Pregnancy
* poorly controlled asthma and cardiovascular disease
* use of drugs that interfere with testing and could not be stopped such as antihistamines, tricyclic antidepressants, antipsychotics, beta blockers, high dose oral glucocorticoids
* Non-IgE mediated type of serious allergic reaction such as Stevens - Johnson syndrome, Toxic Epidermal Necrolysis, and Drug Rash with Eosinophilia and Systemic Symptoms (DRESS) Syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited during the clinical evaluation of labelled penicillin allergy at the regional hospital of Metz, France (Mercy, Centre Hospitalier Régional CHR de Metz - Thioville). All patients were well and had no need of penicillin treatment at the time of evaluation and testing. A detailed history of the probable implicated molecule, the type of the reaction, the age at onset and the received treatment were obtained by Dr SL.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
efficacy of repeated skin testing | week 4
  verified efficacy of repeated skin testing 4 weeks or more after drug provocation test and challenge in distant penicillin allergic patients. The reagents used for skin testing were as follow: Penicillin G, Clamoxyl, Augmentin,Tienam, Histamine and Normal saline (negative control). A skin test producing a papule with a diameter greater then 3 mm is considered as positive.

SECONDARY OUTCOMES:
efficacy of allergy testing | Week 4
  efficacy of allergy testing in identifying penicillin hypersensitivity reactions. Patients were called to perform, once again skin testing because skin tests sooner could result in false negatives due to the temporary desensitized state.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Lefevre, MD, Principal Investigator — CHR Metz Thionville
Locations (1):
- CHR Metz Thionville, Thionville, Moselle, France

IPD SHARING:
Plan to Share IPD: No